CLINICAL TRIAL: NCT05705232
Title: Correlation Between Disease Activity of Inflammatory Bowel Disease, Inflammatory Markers and Peripheral Arthritis .
Brief Title: Inflammatory Marker in Ibd and Peripheral Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mansour Ali, Assistant lecturer, Assiut University
Other Study IDs: IBD and peripheral arthritis
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: IBD-Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Objective Of This Study Is To Estimate The Correlation Between Disease Activity In IBD, Inflammatory Markers And Peripheral Arthritis After Exclusion Of Other Causes Arthritis

DETAILED DESCRIPTION:
Inflammatory Bowel Diseases (IBD) Are Chronic Relapsing Inflammatory Disorder Of The Gastrointestinal Tract (GIT) , Which Represented Mainly By Ulcerative Colitis (UC) And Crohn's Disease .

IBD Is To Be Considered Systemic Disease Since They Are Often Associated With Extra intestinal Manifestation, Especially During Activity, Which Reflect A Pathogenic Mechanism As Arthritis ,Erythema Nodosum ,Pyoderma Gangrenosum , Apthous Ulceration ,Iritis And Uveitis.

Peripheral Arthritis (Pa) Is Observed Rather Than Frequently, The Arthritis Involves Predominantly The Joint Of The Lower Limb ,And In Most Cases It Accompanies The Activity Of The Intestinal Disease Pauciarticular, Asymmetric, Migratory And Non Deforming.

Predicting Relapse By Measuring Non Invasive Biomarkers Could Allow Early Treatment Adaptation .Several Studies Have Shown A Correlation Between Intestinal Inflammation And Serum C-Reactive Protein Or Fecal Calprotectin Levels .

ELIGIBILITY:
Inclusion Criteria:

* 1-Pt Above 18 Yrs. 2- IBD Pt. Confirmed By Colonoscopy 3- IBD Patient with Arthritis During Activity

Exclusion Criteria:

* 1-Age Below 18 Yrs. Old 2-Arthritis Of Other Causes Than IBD PT

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient With inclusion criteria attending Internal Medicine Department clinics ,Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between IBD Patients Presented With Peripheral Arthritis and degree of Disease activity | 1/2/2023to 1/12/2024
  Estimate The Correlation Between Disease Activity In IBD, Inflammatory Markers And Peripheral Arthritis After Exclusion Of Other Causes Arthritis

CONTACTS AND LOCATIONS:
Overall Officials: Eman Mohamed, Study Director — Assiut University; Mostafa Mansor, Principal Investigator — Assiut University; Nabila Fayek, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Palm O, Moum B, Jahnsen J, Gran JT. The prevalence and incidence of peripheral arthritis in patients with inflammatory bowel disease, a prospective population-based study (the IBSEN study). Rheumatology (Oxford). 2001 Nov;40(11):1256-61. doi: 10.1093/rheumatology/40.11.1256. PMID 11709609